CLINICAL TRIAL: NCT04183309
Title: Effects of Pneumoperitoneum on Dynamic Alveolar Stress-strain in Anesthetized Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: 2919/1980/2019
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-02

CONDITIONS: Atelectasis
Keywords: Children; Ultrasound
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric anesthetized patients: Pediatric anesthetized patients undergoing abdominal laparoscopy surgery (simple-arm study).
  Interventions: Other: Measure the transpulmonary pressure in pediatric patients

INTERVENTIONS:
Other: Measure the transpulmonary pressure in pediatric patients — Esophageal pressure will be measured by an esophageal ballon to assess transpulmonary pressure during laparoscopy surgery. Lung collapse will detected when transpulmonary pressure became negative and using lung ultrasound images. Lung ultrasound examinations will be performed at different times-points: after anesthesia induction, 10 minutes after pneumoperitoneum insufflation, and at the end of surgery. A lung recruitment maneuver will be applied if these patients present atelectasis during surgery.

SUMMARY:
General anesthesia is associated with loss of pulmonary functional residual capacity and consequent developement of atelectasis and closure of the small airway. Infants and young children are more susceptible to this lung collapse due to their small functional residual capacity.

Mechanical ventilation in a lung with reduced functional residual capacity and atelectasis increased the dynamic alveolar stress-strain inducing a local inflammatory response in atelectatic lungs areas know as ventilatory induced-lung injury (VILI). This phenomenon may appear even in healthy patients undergoing general anesthesia and predisposes children to hypoxemic episodes that can persist in the early postoperative period. During laparoscopy, pneumoperitoneum may aggravate the reduction of functional residual capacity as it generates a further increase in intra-abdominal pressure.

The increase in alveolar stress-strain cloud be reduced during pneumoperitoneum in theory, if normal functional residual capacity is restored and the transpulmonary pression is reached at the end of expiration of 0-1 cmH2O.

DETAILED DESCRIPTION:
This is a prospective and observational study designed to measure transpulmonary pressure during pneumoperitoneum. The investigators will studied 20 mechanically ventilated pediatric patients schedule for abdominal laparoscopy surgery under general anesthesia.

Lung mechanics will be assessed during laparoscopy. Esophageal pressure will be measured by an esophageal ballon to measure transpulmonary pressure. Lung collapse will detected when transpulmonary pressure became negative and using lung ultrasound images. A lung recruitment maneuver will be applied if these patients present atelectasis during surgery. The optimal level of positive end-expiratory pressure (PEEP) if defined as the PEEP level when transpulmonary pressure remains positive during the PEEP titration trial of the recruitment maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Written Inform Consent by parents
* Programmed surgery
* Laparoscopic surgery
* Supine position
* American Society of Anesthesiologists classification: physical status I-II

Exclusion Criteria:

* Acute airway infection
* Cardiovascular or pulmonary disease

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 3 to 7 years old, schedule for abdominal laparoscopy surgery under general anesthesia with tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Transpulmonary pressure measured by esophageal ballon in pediatric patients | 2 hours
  Effect of pneumoperitoneum on transpulmonary pressure using esophageal ballon in pediatric patients schedule for abdominal laparoscopy surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Tusman, MD, Study Director — Hospital Privado de Comunidad
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No